CLINICAL TRIAL: NCT06245005
Title: Investigation of a Novel Quantitative Measure of Preoperative Cognitive Reserve in Older Surgical Patients: a Feasibility Study
Brief Title: Preoperative Cognitive Reserve in Older Surgical Patients: a Feasibility Study
Status: Recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Michelle Humeidan, Associate Professor, Ohio State University
Other Study IDs: 2022H0419
Record Dates: First submitted 2024-01-18; First posted 2024-02-07 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- OPAC: Feasibility to conduct brain exercise gameplay on a portable electronic device at Ohio State Preoperative Assessment Clinic (OPAC)
  Interventions: Device: Brain exercise gameplay on a portable electronic device
- PREOP: Feasibility to conduct brain exercise gameplay on a portable electronic device at The Wexner Medical Center Preoperative Holding Areas.
  Interventions: Device: Brain exercise gameplay on a portable electronic device

INTERVENTIONS:
Device: Brain exercise gameplay on a portable electronic device — Feasibility is defined as a 70% completion rate for at least 3 of the six brain exercise games in study participants from which a 'first gameplay score' can be determined. Investigators will also assess level of satisfaction with the brain exercise intervention and barriers to playing in the busy preoperative clinical settings as evaluated by a patient-centered questionnaire (Discharge Survey).

SUMMARY:
Investigators will evaluate feasibility of using a custom 6-game Lumosity brain exercise experience in busy clinical areas to obtain a quick, quantitative measure of cognitive reserve (first gameplay performance [FGP]) in older patients presenting for major surgery. Participants in this feasibility trial will serve as a pilot population to estimate postoperative delirium incidence in patients willing and able to complete the brief, self-directed, brain exercise experience on a portable electronic device in various preoperative encounters, and will provide insight into which preoperative encounter (outpatient clinic or morning of surgery preoperative holding) may be more conducive to brief preoperative cognitive evaluations and interventions in future studies. First gameplay performance obtained during study procedures will be compared based upon postoperative delirium status (positive verse negative) to evaluate predictive value of the custom 6-game battery. This will guide future studies of FGP as a quick, quantitative measure of cognitive reserve in older surgical patients, with potentially more utility in preoperative patients than other assessments of cognitive function.

DETAILED DESCRIPTION:
Potential study participants will be identified by researchers monitoring The Ohio State University Preoperative Assessment Clinic (OPAC) and operating room (OR) schedules. Eligible patients will be contacted over-the-phone regarding willingness to participate. Surgeons will be made aware when their patients have been approached over the phone and updated accordingly if the patient agrees to be enrolled in the study. If willing, patients will be met at either their preoperative assessment at OPAC or their day of surgery at Preoperative Holding. Patients will be screened at this encounter for inclusion and exclusion criteria.

Following the initial screening encounter, patients will be required to provide informed consent prior to any study activities or data collection. Once informed consent is signed by both the subject and researcher, the researcher will provide the patient with a portable electronic device (laptop) with access to Lumosity brain exercise software (Lumos Labs, San Francisco, California, USA) and instruct participants to complete as many of the provided 6 games as possible. These 6 games were identified specifically from preliminary data indicating their postoperative delirium predictive capacity. Gameplay completion and performance scores will be coded and stored on the Lumosity software. Personal health information will not be used on the research device.

At this visit, the researcher will also collect demographic information (age, sex, body max index (BMI), ethnicity, and educational level) and relevant comorbidities via the Charlson Comorbidity Index (CCI). The research device will be collected at the end of the patient's visit at OPAC or just prior to surgery when in preoperative holding.

All patients will undergo surgery as planned. Time under anesthesia and type of surgery will be collected. On the first day following surgery, patients will be assessed by research members for the presence of delirium using the 3-Minute Diagnostic Confusion Assessment Method (3D-CAM) at 0800 ± 2 hours and 1700 ± 2 hours. This will be repeated every postoperative day until postoperative day 7 or discharge, whichever comes first. Additionally, medical notes from the day of surgery to discharge or post-operative day (POD) 7 (whichever comes first) will be assessed for delirium by a researcher using a validated medical chart-based delirium assessment (CHART-DEL). Patients will be asked to complete the Discharge Survey Prior to hospital discharge or over the phone after discharge. In addition, their length of stay in the hospital and discharge location will be collected.

ELIGIBILITY:
Inclusion Criteria

1. 60 years of age or older
2. Capable and willing to consent
3. Non-cardiac/non-neurological surgery with an expected hospital stay of at least 72 hours
4. Anticipated ASA physical status I-IV
5. English speaking
6. Willingness to use computer-based device

Exclusion Criteria

1. Severe visual or auditory deficits
2. Illiterate
3. Surgery or procedure within the previous 6 months requiring general anesthesia
4. Active Axis I or II psychiatric disorders including bipolar disorder, schizophrenia, dementia, alcohol, or drug abuse
5. ASA physical status V, VI
6. Planned postoperative ICU admission
7. Preoperative benzodiazepine administration (i.e. Midazolam, Diazepam)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 60 years of age or older, capable and willing to consent and scheduled to undergo non-cardiac/non-neurological surgery with an expected hospital stay of at least 72 hours.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Lumosity 6-game brain exercise completion | up to 30 minutes after participants start the first Lumosity game brain exercise
  Determine if brain exercise gameplay on a portable electronic device is feasible in two different preoperative settings (The Ohio State Preoperative Assessment Clinic (OPAC) and The Wexner Medical Center Preoperative Holding Areas).

SECONDARY OUTCOMES:
Incidence of Postoperative Delirium | through study completion, an average of 7 days
  To assess the incidence of Postoperative Delirium

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
The proportion (95% confidence interval) of patients successfully completing at least three games will be estimated overall and in each setting. Investigators will additionally summarize the total number of games played overall and in each setting. Questionnaire results will be summarized in each setting as absolute data with 0: strongly disagree, 25: disagree, 50: neutral, 75: agree, and 100: strongly agree.